CLINICAL TRIAL: NCT00062049
Title: A Phase I Study of Subcutaneous "CYT 99 007" (Interleukin-7) in Patients With Refractory Non Hematologic Malignancy
Brief Title: Interleukin-7 in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 030152; 03-C-0152I; CDR0000304451; NCT00059059 (obsolete NCT alias)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Interleukin-7

INTERVENTIONS:
Biological: recombinant interleukin-7

SUMMARY:
RATIONALE: Interleukin-7 may stimulate a person's white blood cells to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of interleukin-7 in treating patients with refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and dose-limiting toxicity of biologically active doses of interleukin-7 in patients with refractory solid tumors.
* Determine a range of biologically active doses of this drug in these patients.
* Determine the biological effects of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Determine the antitumor effects of this drug in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive interleukin-7 (IL-7) subcutaneously on days 0, 2, 4, 6, 8, 10, 12, and 14 (for a total of 8 doses) in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of IL-7 until the maximum tolerated dose (MTD) and "biologically active dose" (BAD) are determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The BAD is defined as the dose that produces a sustained 50% increase in CD3+ count over the patient's baseline without unacceptable toxicity.

Patients are followed at 1, 3, and 6 months and at 1 year after study completion.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 3.75-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy meeting both of the following criteria:

  * No known curative therapy
  * Failed standard therapy, defined as either lack of response OR disease progression (i.e., at least 25% increase in disease or new disease)
* Measurable or evaluable disease
* No hematopoietic malignancies
* No primary carcinoma of the lung

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* No proliferative hematologic disease

Hepatic

* AST and ALT less than 3 times upper limit of normal (ULN)
* PT/PTT no greater than 1.5 times ULN
* No documented hepatitis B infection
* No documented hepatitis C infection

Renal

* Creatinine clearance greater than 60 mL/min

Cardiovascular

* Ejection fraction greater than 45% by MUGA
* Hypertension (resting blood pressure greater than 140/90 mm Hg) must be controlled with standard anti-hypertensive therapy

Pulmonary

* No severe asthma
* DLCO/VA greater than 50% of predicted
* FEV_1 greater than 50% of predicted

Immunologic

* No autoimmune disease
* Peripheral CD3+ cell count greater than 300/mm^3 and stable on 4 successive determinations
* HIV negative

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other medical or psychiatric condition that would preclude study compliance
* No cognitive impairment or likelihood of developing cognitive impairment during study participation
* No need for palliative therapy
* No splenomegaly

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy by cytokines, anti-tumor vaccines, or monoclonal antibody therapy prior to the initiation of peripheral CD3 count determination
* No prior allogeneic hematopoietic stem cell transplantation
* No other concurrent immunotherapy
* No other concurrent biologic agents (e.g., growth factors or monoclonal antibodies)

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* No prior systemic corticosteroid therapy for more than 72 hours within the 2 weeks prior to initiation of peripheral CD3 cell count determination
* No concurrent chronic steroid therapy

Radiotherapy

* Not specified

Surgery

* No prior solid organ transplantation
* No prior splenectomy

Other

* More than 4 weeks since prior cytotoxic therapy prior to the initiation of peripheral CD3 cell count determination
* No concurrent cytotoxic therapy
* No concurrent immunosuppressive therapy
* No concurrent medications for the treatment of hypertension
* No concurrent chronic asthma medications
* No concurrent chronic anticoagulants (e.g., high-dose warfarin, heparin, or aspirin)

  * Low-dose oral warfarin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sportes, MD, Study Chair — National Cancer Institute (NCI); Ronald E. Gress, MD — NCI - Experimental Transplantation and Immunology Branch
Locations (3):
- United States (3):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Methodist Hospital, Houston, Texas

REFERENCES:
- [Result] Sportes C, Babb RR, Krumlauf MC, Hakim FT, Steinberg SM, Chow CK, Brown MR, Fleisher TA, Noel P, Maric I, Stetler-Stevenson M, Engel J, Buffet R, Morre M, Amato RJ, Pecora A, Mackall CL, Gress RE. Phase I study of recombinant human interleukin-7 administration in subjects with refractory malignancy. Clin Cancer Res. 2010 Jan 15;16(2):727-35. doi: 10.1158/1078-0432.CCR-09-1303. Epub 2010 Jan 12. PMID 20068111